CLINICAL TRIAL: NCT01030549
Title: Latin American Multicenter Cardiovascular Magnetic Resonance Reference Study
Status: Completed | Type: Observational
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Juliano de Lara Fernandes, Physician Reasearcher, University of Campinas, Brazil
Other Study IDs: CMRLAC-01
Record Dates: First submitted 2009-12-09; First posted 2009-12-11 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
Keywords: cardiovascular magnetic resonance; ventricular volumes; ventricular function; Healthy normal individuals from 20 to 80 years of age

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study was designed to investigate the physiological properties of adult heart using cardiovascular magnetic resonance imaging in normal volunteers in Latin America.

DETAILED DESCRIPTION:
Evaluation of myocardial mass, volumes and function is essential in the management of cardiovascular diseases. While 2D and 3D echocardiography play a major role in determining these parameters cardiovascular magnetic resonance (CMR) has become a widely accepted gold standard for these measurements due to its high accuracy and reproducibility.

However, determining normal reference standards for CMR is crucial for proper use of the method. Previous reports have established normal ranges for both fast low angle shot techniques6 and the more commonly used steady state free precession methods including values normalized not only to body surface area but to age and gender as well. Despite these general references, variability in normal ranges have been reported previously when ethnicity is taken into account. The ongoing Multi-Ethnic Study of Atherosclerosis (MESA) trial has measured cardiovascular function in participants with different ethnical backgrounds, reporting differences in the African-American and Asian-American groups.

Latin-American populations have generally been underrepresented in most clinical cardiovascular trials despite representing a growing percentage of heart disease patients in the world and, particularly, in the USA12-15. While the MESA trial evaluated cardiac function by CMR in Hispanics, data was limited to participants living in USA, within a restricted age group and representing only a small fraction of their entire cohort. It is thus essential to acquire specific data for this population regarding normal CMR values in order to permit not only precise clinical evaluation of Hispanic patients but also accurate assessment of ventricular function figures from Latin American countries in future CMR and drug trials.

To accomplish this goal, we propose a multicenter study to collect CMR data from countries in Latin America in normal participants with 20-80 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic subjects with 20 to 80 years of age with no history of cardiac disease, no known risk factors with normal physical examination and ECG

Exclusion Criteria:

* Current smokers or smokers with < 10 years of quitting
* Systolic blood pressure > 120mmHg or diastolic blood pressure > 80mmHg
* Fasting blood glucose > 100mg/dL
* Total cholesterol > 240mg/dL

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal healthy individuals
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2009-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
CMR data: end-diastolic volume, end-systolic volume, stroke volume, cardiac output, ejection fraction, mass, ascending and descending aortic diameters, aortic arch diameter, atrial diameter, interventricular septum thickness, posterior wall thickness. | At enrollment of patients (time zero). No follow-up will be performed since the trial is cross-sectional

CONTACTS AND LOCATIONS:
Overall Officials: Juliano L Fernandes, MD, PhD, Principal Investigator — University of Campinas, Brazil
Locations (1):
- University of Campinas, Campinas, São Paulo, Brazil